CLINICAL TRIAL: NCT06083376
Title: Effect of Telerehabilitation-based Spinal Stabilization Exercises on Epicardial Adipose Tissue and Exercises Capacity in Individuals With Hypertension
Brief Title: Effect of Spinal Stabilization Exercises on Epicardial Fat Tissue and Exercise Capacity in Hypertensives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Tunç Süygün, LECTURER, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU-TUNCSUYGUN-003
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Epicardial adipose tissue; Hypertension; Exercises Capacity; Telerehabilitation; spinal stabilisation exercise
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental)
  Interventions: Other: Spinal Stabilization Exercise
- control group (Active Comparator)
  Interventions: Other: physical activity counseling

INTERVENTIONS:
Other: Spinal Stabilization Exercise — Spinal stability exercises are commonly used isometric and isotonic exercises. A spinal stabilization exercise training program will be applied to the exercise group participants using the telerehabilitation method (simultaneous connection) 3 days a week for 8 weeks and a total of 24 sessions.
  Arms: exercise group
Other: physical activity counseling — Control group participants will first be given initial evaluations and verbal physical activity recommendations will be given. Patients will be contacted by phone at the 2nd, 4th and 6th weeks and reminded about the importance of physical activity.
  Arms: control group

SUMMARY:
It has been suggested that Epicardial Adipose Tissue (EAT) may be an adjunctive marker to classical risk factors for the presence and severity of coronary artery disease. EAT thickness is also associated with MetS and hypertension, high levels of low-density lipoprotein cholesterol and insulin resistance.Studies have shown that moderate-intensity and high-intensity aerobic exercise and resistance exercise training reduce EAT. However, aerobic and resistance exercises may be found challenging and demanding by individuals and in most cases, high or moderate intensity exercise may be considered difficult. In a study conducted in physically inactive individuals, it was concluded that there was a significant increase in heart rate and BP following spinal stabilisation exercises performed 4 days a week for a total of 8 sessions for 2 weeks, but the increase in these cardiac parameters would tend to decrease following regular exercise. In the current literature, there is no study evaluating the effect of spinal stabilisation exercise on EAT thickness, exercise capacity and cardiovascular parameters in individuals with HT.

Barriers to access to healthcare services such as distance, time and cost can be overcome with technology. COVID-19 has accelerated the transition of many physiotherapy services to telerehabilitation. Evidence has shown that telerehabilitation is an effective delivery model for providing face-to-face physiotherapy services with equal or even superior outcomes, especially in musculoskeletal treatment.

The aim of this study was to determine the effect of spinal stabilisation exercise with telerehabilitation on EAT and exercise capacity in individuals with HT.

ELIGIBILITY:
Inclusion Criteria:

1. Being followed up with Hypertension for at least 6 months
2. Volunteering to participate in the study
3. Speaking Turkish
4. Being literate
5. Not having participated in any structured exercise programme for at least 6 months

Exclusion Criteria:

1. Severe valvular disease
2. Having heart failure
3. Having cardiomyopathy
4. Myocardial infarction at least 6 months ago
5. Stable or unstable angina pectoris
6. Left ventricular ejection fraction below 40
7. Presence of peripheral artery disease
8. History of deep vein thrombosis, pulmonary embolism or stroke in the past
9. Chronic kidney disease
10. Having thyroid diseases
11. Active infectious or inflammatory disease
12. Body Mass Index >40 kg/m2
13. Having a serious psychiatric illness such as panic disorder or major depression

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Change in epicardial fat tissue thickness after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  All patients underwent transthoracic echocardiography conducted by a single cardiologist using a Philips HD11XE (Philips Medical Systems) device in the left lateral decubitus position by the standard technique. Epicardial fat thickness was measured in the parasternal long axis imaging window, using the aortic annulus as an anatomical indicator for vertical measurement, and the widest part of the region from the right ventricular free wall to the pericardium at the end of the systole.
Change in exercises capacity after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  The six-minute walk test (6MWT) will be administered to all participants twice on the same day, half an hour apart. Patients will rest for 10 minutes before the test is performed. Subjects will be asked to walk as fast as possible at their own walking speed for 6 minutes in a 30-meter straight corridor. Every minute during the test, standard phrases will be used to encourage the patient. At the end of the test, 6 minutes walking distance will be recorded. There is no minimum or maximum value as it depends on the person's performance. Longer walking distance indicates better functional capacity.

SECONDARY OUTCOMES:
Change in blood pressure after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Blood pressure and heart rate will be measured with a calibrated digital sphygmomanometer from the calibration unit. Participants will have their blood pressure measured in the morning after taking their current blood pressure medication. Participants will rest in a sitting position for 5 minutes before the measurement. The average of the two SDB and BP measurements will be recorded.
Change in heart rate after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Heart rate will be measured with a calibrated digital sphygmomanometer from the calibration unit. Participants will have their blood pressure measured in the morning after taking their current blood pressure medication. Participants will rest in a sitting position for 5 minutes before the measurement. The average of the two SDB and BP measurements will be recorded.
Change in Evaluation of Spinal Stabilisation Endurance after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  The Bridge Building Test will be used to assess spinal stabilisation endurance. Participants were asked to lift their hips off the bed in the supine position and maintain the position without breaking the position. The time they maintain the position will be recorded in seconds.
Evaluation of Stabilisation Strength of Deep Spinal Muscles after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Stabilisation ability of deep spinal muscles will be evaluated by using "The Stabilizer Pressure Biofeedback Unit" (BGU). The BGU is a device designed by physiotherapists that shows the pressure change in a cell that is filled with air and pressurised. The stabiliser is used to monitor, measure and provide feedback on the movement of the relevant body segment. During the test, participants are asked to lie face down with their head turned to one side. The three-chamber pressure cell of the device is placed in the lower part of the abdominal region and in the centre of the spina iliaca anterior superior. Once the pressure of the manometer is inflated to 70 mmHg, the participants are asked to pull the abdominal wall inwards without any spinal or pelvic movement, as previously taught. Pressure readings for measurement are taken 3 times in succession for 10 seconds.
Evaluation of Peripheral Muscle Strength after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  5 repetition sit and stand test (5TOKT): It is a performance test in which dynamic balance is evaluated by recording the performance of the individuals to sit and stand on a chair 5 times serially in terms of time. To measure the 5TOKT time, the participants are asked to sit on a chair that is not fixed to the floor, without armrests, 45 cm high, with a flat back and a hard floor, with their backs touching the back of the chair and their hands crossed in front of their torso. The participants sit on and off the chair 5 times as fast as they can following the 'Go' command of the assessor
Evaluation of Peripheral Muscle Strength after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Hand grip strength will be evaluated with a hand dynamometer (Saehan hydraulic dynamometer). The measurement will be made in the dominant hand. Grip strength measurements for the dominant hand of the volunteers will be taken three times and the highest value in kilograms (kg) will be recorded for statistical evaluation. There will be a break of at least one minute between each trial.
Evaluation of functional mobility and balance after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  The Time Up and Go Test (TUG) will be used to measure functional mobility and balance in individuals. It is a practical method that does not require equipment. During the test, the participant sits in the chair at the beginning, gets up from the chair with the start command, goes to the place marked 3 m ahead, returns and sits back in the chair. The time is recorded in seconds
Evaluation of Quality of Life after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  The EQ-5D Quality of Life Scale will be used to assess the quality of life of the participants. It consists of five dimensions including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The answers to each dimension have 3 options: no problem, some problem and major problem. The index values of the scale are calculated on the computer using an excel format prepared by the Euro Quality of Life group based on formulae calculated from different population samples. The answers obtained from these patients are placed on this programme.
  It is the calculation of individual-specific index values ranging between 0 and 1. In index scores, a value of 0 indicates death and a value of 1 indicates perfect health. The scale developers did not specify minimum and maximum values.
Evaluation of healthy life profile after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Healthy life profile will be evaluated with the Healthy Lifestyle Behaviours Scale. The scale was developed by Walker et al. The scale was revised in 1996 and named as Healthy Lifestyle Behaviours Scale-II. The Turkish validity and reliability study was conducted by Bahar et al. in 2008. The scale has 52 items and consists of six factors. These are health responsibility, physical activity, nutrition, spiritual development, interpersonal relationships and stress management. The scale rating is in 4-point Likert type. Never (1), sometimes (2), frequently (3) and regularly (4) are accepted. The lowest score that can be obtained from the whole scale is 52 and the highest score is 208.
Evaluation of Activity of Daily Living after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Nottingham Extended Activities of Daily Living (NADL) for assessing GYA Index (NGGYA) will be used. It consists of 22 questions. All questions are answered on a scale from 0 to 3 points. It has 4 subscales; movement, in the kitchen, housework, leisure activities. The sum of these 4 subscales gives the total score. The highest possible score is 66. Turkish validity and reliability study was conducted by Şahin et al.
Evaluation of Activity of Physical Activity after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Physical activity level was evaluated with the Turkish version of the International Physical Activity Questionnaire-7, whose reliability and validity. The International Physical Activity Questionnaire-7 is a seven-item questionnaire that assesses severe physical activity (duration: min and frequency: day), moderate physical activity (duration: min and frequency: day), and walking time of at least 10 minutes (frequency: day) over the previous seven days. The metabolic equivalent of task (MET) corresponding to the basal metabolic rate is converted from severe and moderate activity and walking periods, and the overall physical activity score (MET- min/week) is determined. Higher scores indicate higher levels of physical activity. There is no minimum or maximum value since it depends on performance in daily life.
Evaluation of Self-Efficacy and Self-Management after 8 weeks-24 sessions of exercise | baseline and 8 weeks
  Heart Health Self-Efficacy and Self-Management Scale was developed by Maria Mares et al. It is a 12-item scale that can evaluate the concepts of self-efficacy and self-effectiveness, which are prominent in disease management. Both English and Arabic languages were used in the scale development study. Turkish adaptation study (Karamanoğlu Mehmetbey University Faculty of Medicine Ethics Committee Decision No 04-202l/04) Süygün et al. A minimum of 0 and a maximum of 48 points can be obtained. Higher scores indicate better self-efficacy and self-management.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoğlu Mehmetbey University, Merkez, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Tunc Suygun E, Suygun H, Senalp ZE, Vardar Yagli N. The effect of telerehabilitation-based core stabilization exercises on epicardial fat tissue and exercise capacity in hypertensives. Disabil Rehabil. 2025 Nov 24:1-12. doi: 10.1080/09638288.2025.2593190. Online ahead of print. PMID 41283774